CLINICAL TRIAL: NCT02258451
Title: A Phase II Randomized, Double-blind, Placebo-controlled Trial of Radium-223 Dichloride in Combination With Exemestane and Everolimus Versus Placebo in Combination With Exemestane and Everolimus When Administered to Metastatic HER2 Negative Hormone Receptor Positive Breast Cancer Subjects With Bone Metastases
Brief Title: Study of Radium-223 Dichloride in Combination With Exemestane and Everolimus Versus Placebo in Combination With Exemestane and Everolimus in Subjects With Bone Predominant HER2 Negative Hormone Receptor Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17096; 2014-002114-23 (EudraCT Number)
Record Dates: First submitted 2014-09-30; First posted 2014-10-07 (Estimated); Results first posted 2022-03-10 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — radium Ra 223 dichloride; Sodium Chloride; exemestane; Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radium-223 dichloride + exemestane/everolimus (Experimental): Up to 6 cycles of radium-223 dichloride 50kBq/kg body weight (55 kBq/kg after implementation of National Institute of Standards and Technology [NIST] update) (randomized). Participants will also receive exemestane, 25-mg tablet once daily (after a meal), and everolimus, 10 mg once daily (with or without food), and supportive care as per the local or institutional standard of practice.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Exemestane; Drug: Everolimus
- Placebo + exemestane/everolimus (Placebo Comparator): Up to 6 cycles of saline injection (placebo) (randomized). Participants will also receive exemestane, 25-mg tablet once daily (after a meal), and everolimus, 10 mg once daily (with or without food), and supportive care as per the local or institutional standard of practice.
  Interventions: Drug: Placebo (saline); Drug: Exemestane; Drug: Everolimus

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Up to 6 cycles of radium-223 dichloride 50kBq/kg body (55 kBq/kg after implementation of NIST update)
  Arms: Radium-223 dichloride + exemestane/everolimus
Drug: Placebo (saline) — Up to 6 cycles of saline injection
  Arms: Placebo + exemestane/everolimus
Drug: Exemestane — One 25 mg tablet once daily after a meal.
Drug: Everolimus — The recommended dose of everolimus administered in the study is 10 mg once daily with or without food.
  Starting dose, dose modifications, and administration of exemestane and everolimus must be in compliance with the local labels in each of the participating countries and/or in line with local standard of practice.

SUMMARY:
The objective of this study is to assess efficacy and safety of radium 223 dichloride in subjects with human epidermal growth factor receptor 2 (HER2) negative hormone receptor positive breast cancer with bone metastases treated with exemestane and everolimus

After implementation of CSP Amendment 10, only a limited number of subjects will remain in this study, in order to reduce the burden to study subjects, collection of data will be reduced and will focus mainly on acute safety, SSE, and OS. Once subjects are rolled over, the long-term safety will be collected and assessed entirely in the separate extended safety follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Women (≥18 years of age) with metastatic breast cancer not amenable to curative treatment by surgery or radiotherapy.
* Documentation of histological or cytological confirmation of estrogen receptor positive (ER+) and HER2 negative adenocarcinoma of the breast must be available.
* Documentation of menopausal status: postmenopausal subjects or pre-menopausal subjects with ovarian radiation or concomitant therapy with a luteinizing hormone-releasing hormone (LH-RH) agonist/antagonist are eligible.
* Subjects with bone dominant disease with at least 2 skeletal metastases identified at baseline by bone scintigraphy and confirmed by computed tomography (CT)/magnetic resonance imaging (MRI).
* Subjects must have received at least one line of hormonal therapy in the metastatic setting.
* Subjects who are eligible as per the Investigator's assessment and according to the local label for treatment with exemestane and everolimus as a second line or greater of hormone therapy in a metastatic setting.
* Subjects must have experienced recurrent/progressive disease following treatment with a non-steroidal aromatase inhibitor (letrozole or anastrozole) in an adjuvant or metastatic setting
* Subjects must have experienced no more than two skeletal-related events (SREs) prior to study entry defined as: need for external beam radiotherapy (EBRT) to bone pain, pathological bone fracture (excluding major trauma), spinal cord compression and/or orthopedic surgical procedure. Subjects with no prior SREs are not permitted.
* Subjects must be on therapy with bisphosphonates or denosumab for at least 1 month before start of study treatment.
* Adequate hematological, liver and kidney function.

Exclusion Criteria:

* Subjects with Inflammatory breast cancer.
* Patients with immediately life-threatening visceral disease for whom chemotherapy is preferred treatment option.
* Subjects who have either received chemotherapy for metastatic disease or are considered by the treating investigator to be appropriate candidates for chemotherapy as current treatment for metastatic breast cancer are excluded. Chemotherapy administered for adjuvant/neo adjuvant disease is acceptable provided it was administered at least 1 year prior to study entry.
* Subjects who received prior treatment or are already receiving everolimus treatment prior to study entry are not eligible.
* Subjects with known or history of brain metastases or leptomeningeal disease: subjects with neurological symptoms must undergo a contrast CT scan or MRI of the brain within 28 days prior to randomization to exclude active brain metastasis. Imaging of the central nervous system (CNS) is otherwise not required.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (81):
- United States (15):
  - La Jolla, California
  - Los Angeles, California
  - New Haven, Connecticut
  - Hollywood, Florida
  - Ashland, Kentucky
  - Rockville, Maryland
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Pontiac, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Newark, New Jersey
  - Jamaica, New York
  - Watertown, South Dakota
  - Spokane, Washington
- Innsbruck, Austria
- Belgium (4):
  - Brussels
  - Edegem
  - Kortrijk
  - Leuven
- France (5):
  - Angers
  - Nantes
  - Nîmes
  - Saint-Cloud
  - Tours
- Herne, North Rhine-Westphalia, Germany
- Hong Kong (3):
  - Chai Wan
  - Hong Kong
  - Kowloon
- Israel (8):
  - Afula
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
  - Zrifin
- Italy (9):
  - Bari, Apulia
  - Bologna, Emilia-Romagna
  - Forlì Cesena, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Cremona, Lombardy
  - Milan, Lombardy
  - Pisa, Tuscany
- Japan (8):
  - Nagoya, Aichi-ken
  - Sapporo, Hokkaido
  - Sayama, Osaka
  - Hidaka, Saitama
  - Kita-Adachigun, Saitama
  - Koto-ku, Tokyo
  - Kagoshima
  - Osaka
- Oslo, Norway
- Poland (5):
  - Bialystok
  - Gdansk
  - Gdynia
  - Poznan
  - Warsaw
- Singapore, Singapore
- South Korea (6):
  - Suwon, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Daegu
  - Incheon
  - Seoul
- Spain (5):
  - Palma de Mallorca, Illes Baleares
  - Barcelona
  - Madrid
  - Pamplona
  - Seville
- Aarau, Canton of Aargau, Switzerland
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- United Kingdom (5):
  - Truro, Cornwall
  - Plymouth, Devon
  - Nottingham, Nottinghamshire
  - Taunton, Somerset
  - Bristol

REFERENCES:
- [Derived] Rugo HS, Van Poznak CH, Neven P, Danielewicz I, Lee SC, Campone M, Chik JYK, Vega Alonso E, Naume B, Brain E, Siegel JM, Li R, Uema D, Wagner VJ, Coleman RE. Radium-223 in women with hormone receptor-positive bone-metastatic breast cancer receiving endocrine therapy: pooled analysis of two international, phase 2, randomized, double-blind, placebo-controlled trials. Breast Cancer Res Treat. 2024 Apr;204(2):249-259. doi: 10.1007/s10549-023-07147-z. Epub 2023 Dec 20. PMID 38123789
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/17096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted with first participant first visit on 04-JUN-2015 and last participant last visit on 28-OCT-2022.
Pre-assignment Details: Overall, 389 participants were screened and 283 were assigned to treatment. Of these, 142 in the radium 223 dichloride arm and 141 in the placebo arm.
Groups:
- Radium-223 + EXE/EVE: Participants randomized to treatment with radium-223 dichloride, 50 kBq/kg body weight (55 kBq/kg after implementation of NIST update) also received exemestane (EXE), 25-mg tablet once daily (after a meal), and everolimus (EVE), 10 mg once daily (with or without food), and supportive care as per the local or institutional standard of practice
- Placebo + EXE/EVE: Participants randomized to treatment with placebo, also received exemestane (EXE), 25-mg tablet once daily (after a meal), and everolimus (EVE), 10 mg once daily (with or without food), and supportive care as per the local or institutional standard of practice
Period: Overall Study
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Started (Randomized) | 142 | 141
Completed (As exemestane and everolimus given in this study as study treatment was of indefinite duration and ended only at progression, withdrawal, death, or study termination, no participants were considered to have completed their respective treatment regimen. However, all participants discontinued all study treatments.) | 0 | 0
Not Completed | 142 | 141
Not completed — Discontinuation all treatment due to progressive disease - radiological progression | 90 | 101
Not completed — Discontinuation all treatment due to progressive disease - clinical progression | 7 | 7
Not completed — Discontinuation all treatment due to adverse event not associated with clinical disease progression | 8 | 1
Not completed — Discontinuation all treatment due to adverse event associated with clinical disease progression | 8 | 6
Not completed — Discontinuation all treatment due to death | 4 | 3
Not completed — Discontinuation all treatment due to withdrawal by participant | 21 | 13
Not completed — Discontinuation all treatment due to end point reached | 1 | 1
Not completed — Discontinuation all treatment due to physician decision | 0 | 2
Not completed — Discontinuation all treatment due to study terminated by sponsor | 0 | 3
Not completed — Other reason | 1 | 1
Not completed — Never treated | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Analysis Set (ITT analysis set): included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE | Total
Number analyzed (Participants) | 142 | 141 | 283
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.95 (10.40) | 59.08 (11.64) | 59.52 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 141 | 283
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 127 | 125 | 252
  Unknown or Not Reported | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Skeletal Event-free Survival (SSE-FS)
Description: Time from date of randomization to occurrence of one of the following, whichever happened earlier: 1) an on study SSE, which was defined as the use of external beam radiotherapy (EBRT) to relieve skeletal symptoms, the occurrence of new symptomatic pathological bone fractures (vertebral or nonvertebral), the occurrence of spinal cord compression, a tumor related orthopedic surgical intervention; or 2) death from any cause. Per Protocol Amendment 10, following primary analysis completion, further assessments were focused on safety, and only limited efficacy data including SSE and survival were collected and not designed to support reconsideration of the primary analysis efficacy conclusions. Accordingly, no formal statistical analyses were performed for primary and secondary efficacy outcomes in the final analysis. All primary and secondary efficacy outcome measures presented in this document came from the primary completion analysis.
Time Frame: Up to 55 months
Population: Intent to treat analysis set: all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 142 | 141
Months | 21.1 [17.1 to 23.6] | 19.9 [16.2 to 24.2]
Statistical Analysis 1: Comparison: Radium-223 + EXE/EVE vs Placebo + EXE/EVE; The 1-sided null hypothesis that treatment with radium-223 dichloride does not result in superior SSE-FS to treatment with placebo in participant population was tested against the 1-sided alternative hypothesis that the treatment with radium-223 dichloride results in superior SSE-FS time to treatment the placebo. H0: SSE-FS Radium-223+Exemestane/Everolimus <= SSE-FS Placebo+Exemestane/Everolimus, versus HA: SSE-FSRadium-223+Exemestane/Everolimus > SSE-FS Placebo+Exemestane/Everolimus; Test type: Superiority; p = 0.4843, Log Rank — 1-sided SSE-FS hypotheses were tested using a log-rank test with a 2-sided alpha of 0.2, stratified by the randomization stratification factors; Hazard Ratio (HR) = 0.891, 80% CI 2-sided [0.720 to 1.102] — The hazard ratio (radium-223 dichloride / placebo) for SSE-FS was calculated using Cox Proportional Hazards Model, stratified by the same stratification factors as randomization

2. Secondary Outcome: Overall Survival
Description: The time from the date of randomization to the date of death due to any cause. Per Protocol Amendment 10, following primary analysis completion, further assessments were focused on safety, and only limited efficacy data including SSE and survival were collected and not designed to support reconsideration of the primary analysis efficacy conclusions. Accordingly, no formal statistical analyses were performed for primary and secondary efficacy outcomes in the final analysis. All primary and secondary efficacy outcome measures presented in this document came from the primary completion analysis.
Time Frame: Up to 55 months
Population: Intent to treat analysis set: all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 142 | 141
Months | 25.0 [23.0 to 31.4] | 26.4 [21.7 to 28.9]
Statistical Analysis 1: Comparison: Radium-223 + EXE/EVE vs Placebo + EXE/EVE; Test type: Superiority; p = 0.8438, Log Rank — P-value was calculated using a 2-sided log-rank test stratified by the same stratification factors as randomization. No alpha adjustment for multiplicity was applied; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.697 to 1.343] — The hazard ratio (radium-223 dichloride / placebo) was calculated using Cox Proportional Hazards Model , stratified by the same stratification factors as randomization

3. Secondary Outcome: Time to Opiate Use for Cancer Pain
Description: Interval from the date of randomization to the date of opiate use
Time Frame: Up to 55 months
Population: Safety analysis set: all randomized participants who received at least one dose of any study medication (radium 223 dichloride or placebo, exemestane, and everolimus). Participants were assigned to the Radium-223 dichloride arm if they received any dose of Radium-223 dichloride, otherwise to the placebo arm.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Radium-223 + EXE/EVE: Participants who received treatment with radium-223 dichloride, 50 kBq/kg body weight (55 kBq/kg after implementation of NIST update) also received exemestane (EXE), 25-mg tablet once daily (after a meal), and everolimus (EVE), 10 mg once daily (with or without food), and supportive care as per the local or institutional standard of practice
- Placebo + EXE/EVE: Participants did not receive any radium-223 dichloride, but received treatment with any study treatment (placebo, exemestane [25-mg tablet once daily (after a meal)], and everolimus [10 mg once daily (with or without food)]), and supportive care as per the local or institutional standard of practice
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Months | 21.4 [13.2 to NA] — N/A = Value cannot be estimated due to censored data. Insufficient number of participants with events. | 18.4 [8.3 to NA] — N/A = Value cannot be estimated due to censored data. Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Radium-223 + EXE/EVE vs Placebo + EXE/EVE; Test type: Superiority; p = 0.8811, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.962, 95% CI 2-sided [0.577 to 1.604] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Time to Pain Progression
Description: Time from randomization to the first date a participant experienced pain progression based on WPS. Pain progression was defined as an increase of 2 or more points in the BPI-SF "Worst pain in 24 hours" score from baseline observed at 2 consecutive evaluations ≥4 weeks apart or an increase in pain management (IPM) with respect to baseline, whichever occurred first. An IPM is defined as the initiation of any opioid in participants not taking opioids at baseline, the initiation of a strong opioid in participants taking a weak opioid at baseline, or the initiation of an additional strong opioid in participants taking a strong opioid at baseline.
Time Frame: Up to 55 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Months | 7.6 [6.2 to 13.2] | 5.7 [4.9 to 8.5]
Statistical Analysis 1: Comparison: Radium-223 + EXE/EVE vs Placebo + EXE/EVE; Participants with baseline WPS > 8 were included in the analysis population but censored at Day 1; Test type: Superiority; p = 0.6537, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.928, 95% CI 2-sided [0.667 to 1.289] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Time to Cytotoxic Chemotherapy
Description: Time from the date of randomization to the date of the first cytotoxic chemotherapy
Time Frame: Up to 55 months
Population: ITT analysis set: included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 142 | 141
Months | 13.7 [9.9 to 15.8] | 11.6 [9.0 to 16.4]
Statistical Analysis 1: Comparison: Radium-223 + EXE/EVE vs Placebo + EXE/EVE; Test type: Superiority; p = 0.4496, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.884, 95% CI 2-sided [0.641 to 1.219] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Radiological Progression-free Survival (rPFS)
Description: Time from the date of randomization to the date of confirmed radiological progression in either soft tissue, viscera or bone, or death (if death occurs before progression). Progression is defined using the modified RECIST 1.1 criteria (the modification refers to bone lesions assessment). Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or an unequivocal increase in non-target lesions, or the appearance of new lesions. All bone lesions are considered non-measurable and new bone lesions identified by bone scan should be confirmed by further imaging (CT/MRI). If a new bone lesion or unequivocal increase in size of bone lesions is only visible on a CT/MRI and not visible on a technetium-99m bone scan, progression should be declared without further confirmation.
Time Frame: Up to 55 months
Population: ITT analysis set: included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 142 | 141
Months | 7.9 [6.2 to 9.7] | 6.7 [5.4 to 8.1]
Statistical Analysis 1: Comparison: Radium-223 + EXE/EVE vs Placebo + EXE/EVE; Test type: Superiority; p = 0.3467, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.874, 95% CI 2-sided [0.660 to 1.157] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Percentage of Participants With Pain Improvement
Description: In the percentage of participants with confirmed pain improvement. Confirmed pain improvement is defined a 2-point decrease or more in BPI-SF WPS from baseline over 2 consecutive measurements conducted at least 4 weeks apart, without an increase in pain management (IPM). An IPM is defined as the initiation of any opioid in participants not taking opioids at baseline, the initiation of a strong opioid in participants taking a weak opioid at baseline, or the initiation of an additional strong opioid in participants taking a strong opioid at baseline.
Time Frame: Up to 55 months
Population: Safety analysis set with baseline WPS >= 2: all randomized participants who received at least one dose of any study medication (radium 223 dichloride or placebo exemestane, or everolimus), and who in addition had baseline BPI-SF WPS >= 2. Participants were assigned to the Radium-223 dichloride arm if they received any dose of Radium-223 dichloride, otherwise to the placebo arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 91 | 96
percentage of participants | 38.5 [28.4 to 49.2] | 34.4 [25.0 to 44.8]
Statistical Analysis 1: Comparison: Radium-223 + EXE/EVE vs Placebo + EXE/EVE; Test type: Superiority; p = 0.556, Cochran-Mantel-Haenszel — P-value was calculated using a 2-sided Cochran-Mantel-Haenszel test stratified by the same stratification factors as randomization. No alpha adjustment for multiplicity was applied; Risk Difference (RD) = 4.1, 95% CI 2-sided [-10.2 to 18.4]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence (i.e. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation participant after providing written informed consent for participation in the study. AEs were considered to be treatment-emergent if they started or worsened after first application of study intervention up to 30 days after end of treatment with study intervention. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly; another medical important serious event as judged by the investigator and an occurrence of any additional malignancies, including acute myelocytic leukemia or hematological conditions.
Time Frame: From first dosing up to 30 days after the last administration of study treatments, up to 72.6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Participants
  Any TEAE | 139 | 136
  Serious TEAE | 57 | 55
  Radium-223/Placebo-related TEAEs | 73 | 50
  Exemestane-related TEAEs | 75 | 64
  Everolimus-related TEAEs | 130 | 125

9. Secondary Outcome: Number of Participants With Post-treatment Chemotherapy Related Adverse Events
Description: According to protocol amendment 10, all participants who completed the EOT visit will be transferred to a separate extended safety follow-up study for their remaining follow-up. Thus, no further post-treatment data were collected after protocol amendment 10.
Time Frame: From post-treatment till end of study, up to 45.8 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Participants
  All system organ classes_Any_Grade 3 | 1 | 0
  All system organ classes_Any_Grade 4 | 1 | 0
  Blood and lymphatic system disorders_Any_Grade 3 | 1 | 0
  Blood and lymphatic system disorders_Febrile neutropenia_Grade 3 | 1 | 0
  Investigations_Any_Grade 4 | 1 | 0
  Investigations_Neutrophil count decreased_Grade 4 | 1 | 0

10. Secondary Outcome: Number of Participants With Hematological Toxicities: Worst Grade Under Treatment
Time Frame: From first dosing up to 30 days after the last administration of study treatments, up to 72.6 months
Population: Safety analysis set with at least one hematology lab assessment: all randomized participants who received at least one dose of any study medication (radium 223 dichloride or placebo, exemestane, and everolimus), and who in addition had at least one hematology lab assessment. Participants were assigned to the Radium-223 dichloride arm if they received any dose of Radium-223 dichloride, otherwise to the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 137
Participants
  Anemia: Grade 1 | 61 | 57
  Anemia: Grade 2 | 43 | 55
  Anemia: Grade 3 | 21 | 11
  Anemia: Grade 4 | 0 | 0
  Anemia: Normal | 14 | 14
  Leukocytosis: Grade 1 | 0 | 0
  Leukocytosis: Grade 2 | 0 | 0
  Leukocytosis: Grade 3 | 0 | 0
  Leukocytosis: Grade 4 | 0 | 0
  Leukocytosis: Normal | 139 | 137
  Hemoglobin increased: Grade 1 | 0 | 0
  Hemoglobin increased: Grade 2 | 1 | 0
  Hemoglobin increased: Grade 3 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0
  Hemoglobin increased: Normal | 138 | 137
  Lymphocyte count decreased: Grade 1 | 20 | 33
  Lymphocyte count decreased: Grade 2 | 63 | 45
  Lymphocyte count decreased: Grade 3 | 43 | 24
  Lymphocyte count decreased: Grade 4 | 2 | 0
  Lymphocyte count decreased: Normal | 11 | 35
  Lymphocyte count increased: Grade 1 | 0 | 0
  Lymphocyte count increased: Grade 2 | 2 | 2
  Lymphocyte count increased: Grade 3 | 0 | 0
  Lymphocyte count increased: Grade 4 | 0 | 0
  Lymphocyte count increased: Normal | 137 | 135
  Neutrophil count decreased: Grade 1 | 23 | 30
  Neutrophil count decreased: Grade 2 | 48 | 28
  Neutrophil count decreased: Grade 3 | 19 | 0
  Neutrophil count decreased: Grade 4 | 0 | 2
  Neutrophil count decreased: Normal | 49 | 77
  Platelet count decreased: Grade 1 | 60 | 60
  Platelet count decreased: Grade 2 | 7 | 3
  Platelet count decreased: Grade 3 | 7 | 0
  Platelet count decreased: Grade 4 | 1 | 0
  Platelet count decreased: Normal | 64 | 74
  White blood cell decreased: Grade 1 | 37 | 48
  White blood cell decreased: Grade 2 | 59 | 37
  White blood cell decreased: Grade 3 | 17 | 3
  White blood cell decreased: Grade 4 | 1 | 1
  White blood cell decreased: Normal | 25 | 48

11. Secondary Outcome: Number of Participants With New Primary Malignancies
Time Frame: From first dosing till end of study, up to 72.6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Participants | 1 | 0

12. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (From First Dosing Till Primary Analysis)
Description: as for outcome 8
Time Frame: From first dosing till primary analysis cutoff date, up to 55 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Participants
  Any TEAE | 139 | 136
  Serious TEAE | 57 | 53
  Radium-223/Placebo-related TEAEs | 73 | 50
  Exemestane-related TEAEs | 75 | 64
  Everolimus-related TEAEs | 130 | 125

13. Other Pre Specified Outcome: Number of Participants With Post-treatment Chemotherapy Related Adverse Events (From First Dosing Till Primary Analysis)
Time Frame: From post-treatment till primary analysis cutoff date, up to 55 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Participants
  All system organ classes_Any_Grade 3 | 1 | 0
  All system organ classes_Any_Grade 4 | 1 | 0
  Blood and lymphatic system disorders_Any_Grade 3 | 1 | 0
  Blood and lymphatic system disorders_Febrile neutropenia_Grade 3 | 1 | 0
  Investigations_Any_Grade 4 | 1 | 0
  Investigations_Neutrophil count decreased_Grade 4 | 1 | 0

14. Other Pre Specified Outcome: Number of Participants With Hematological Toxicities: Worst Grade Under Treatment (From First Dosing Till Primary Analysis)
Time Frame: From first dosing till primary analysis cutoff date, up to 55 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 137
Participants
  Anemia: Grade 1 | 61 | 57
  Anemia: Grade 2 | 43 | 55
  Anemia: Grade 3 | 21 | 11
  Anemia: Grade 4 | 0 | 0
  Anemia: Normal | 14 | 14
  Leukocytosis: Grade 1 | 0 | 0
  Leukocytosis: Grade 2 | 0 | 0
  Leukocytosis: Grade 3 | 0 | 0
  Leukocytosis: Grade 4 | 0 | 0
  Leukocytosis: Normal | 139 | 137
  Hemoglobin increased: Grade 1 | 0 | 0
  Hemoglobin increased: Grade 2 | 1 | 0
  Hemoglobin increased: Grade 3 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0
  Hemoglobin increased: Normal | 138 | 137
  Lymphocyte count decreased: Grade 1 | 20 | 33
  Lymphocyte count decreased: Grade 2 | 63 | 45
  Lymphocyte count decreased: Grade 3 | 43 | 24
  Lymphocyte count decreased: Grade 4 | 2 | 0
  Lymphocyte count decreased: Normal | 11 | 35
  Lymphocyte count increased: Grade 1 | 0 | 0
  Lymphocyte count increased: Grade 2 | 2 | 2
  Lymphocyte count increased: Grade 3 | 0 | 0
  Lymphocyte count increased: Grade 4 | 0 | 0
  Lymphocyte count increased: Normal | 137 | 135
  Neutrophil count decreased: Grade 1 | 24 | 29
  Neutrophil count decreased: Grade 2 | 47 | 28
  Neutrophil count decreased: Grade 3 | 19 | 0
  Neutrophil count decreased: Grade 4 | 0 | 2
  Neutrophil count decreased: Normal | 49 | 78
  Platelet count decreased: Grade 1 | 60 | 61
  Platelet count decreased: Grade 2 | 7 | 2
  Platelet count decreased: Grade 3 | 7 | 0
  Platelet count decreased: Grade 4 | 1 | 0
  Platelet count decreased: Normal | 64 | 74
  White blood cell decreased: Grade 1 | 37 | 47
  White blood cell decreased: Grade 2 | 59 | 36
  White blood cell decreased: Grade 3 | 17 | 3
  White blood cell decreased: Grade 4 | 1 | 1
  White blood cell decreased: Normal | 25 | 50

15. Other Pre Specified Outcome: Number of Participants With New Primary Malignancies During Study Treatment Till Primary Analysis
Time Frame: From first dosing till primary analysis cutoff date, up to 55 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
Number analyzed (Participants) | 139 | 139
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Time Frame for AE: After providing written informed consent for participation in the study till end of study, up to 73.5 months. Time Frame for the all-cause mortality: Considers all deaths that occurred at any time during the study of 17096 before the last contact, up to 73.5 months.
Description: For All-Cause Mortality section, "Total Number Affected" are updated in final results posting. Deaths of this study 17096 participants who transferred to study 16996 (NCT02312960) for long-term follow-up were erroneously reported in the 17096 primary analysis disclosure. This has been corrected and only 17096 data is reported in this disclosure here. 16996 outcomes will be reported in the 16996 disclosure.
Groups:
- Radium-223 + EXE/EVE: Participants were randomized to treatment with radium-223 dichloride, also with exemestane and everolimus and supportive care as per the local or institutional standard of practice
- Placebo + EXE/EVE: Participants were randomized to treatment with placebo, also with exemestane and everolimus and supportive care as per the local or institutional standard of practice
Arm/Group | Radium-223 + EXE/EVE | Placebo + EXE/EVE
All-Cause Mortality (participants affected / at risk) | 66/139 | 67/139
Serious Adverse Events (participants affected / at risk) | 61/139 | 56/139
Other Adverse Events (participants affected / at risk) | 139/139 | 135/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 + EXE/EVE (N=139) | Placebo + EXE/EVE (N=139)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 5 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Death (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (5)
Sudden death (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (2)
General physical health deterioration (General disorders) | 2 (3) | 3 (4)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 4 (5)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (2)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1)
Biopsy lung (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Appendix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysmetria (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (3)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0)
Medullary compression syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (3) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 + EXE/EVE (N=139) | Placebo + EXE/EVE (N=139)
Anaemia (Blood and lymphatic system disorders) | 55 (191) | 40 (146)
Leukopenia (Blood and lymphatic system disorders) | 12 (49) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 29 (73) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (58) | 9 (19)
Vertigo (Ear and labyrinth disorders) | 8 (10) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 11 (13)
Abdominal pain upper (Gastrointestinal disorders) | 15 (18) | 7 (8)
Constipation (Gastrointestinal disorders) | 6 (7) | 20 (23)
Diarrhoea (Gastrointestinal disorders) | 42 (66) | 31 (54)
Dry mouth (Gastrointestinal disorders) | 10 (13) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 7 (8)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 10 (19)
Nausea (Gastrointestinal disorders) | 41 (55) | 30 (42)
Stomatitis (Gastrointestinal disorders) | 66 (144) | 69 (172)
Vomiting (Gastrointestinal disorders) | 25 (32) | 22 (31)
Asthenia (General disorders) | 29 (48) | 26 (52)
Fatigue (General disorders) | 38 (66) | 41 (60)
Oedema peripheral (General disorders) | 26 (37) | 25 (34)
Pyrexia (General disorders) | 20 (27) | 13 (16)
Peripheral swelling (General disorders) | 8 (8) | 10 (17)
Conjunctivitis (Infections and infestations) | 8 (8) | 3 (3)
Cystitis (Infections and infestations) | 4 (4) | 7 (8)
Nasopharyngitis (Infections and infestations) | 7 (7) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 15 (22) | 20 (38)
Urinary tract infection (Infections and infestations) | 12 (16) | 12 (14)
Alanine aminotransferase increased (Investigations) | 21 (51) | 23 (52)
Aspartate aminotransferase increased (Investigations) | 19 (44) | 21 (40)
Blood cholesterol increased (Investigations) | 15 (22) | 10 (22)
Blood creatinine increased (Investigations) | 11 (26) | 10 (23)
Lymphocyte count decreased (Investigations) | 8 (36) | 7 (14)
Neutrophil count decreased (Investigations) | 14 (43) | 6 (11)
Platelet count decreased (Investigations) | 12 (42) | 12 (28)
Weight decreased (Investigations) | 28 (37) | 22 (31)
White blood cell count decreased (Investigations) | 13 (43) | 13 (31)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 (28) | 6 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (36) | 18 (41)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 (29) | 11 (38)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 8 (14)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (29) | 14 (27)
Hypophosphataemia (Metabolism and nutrition disorders) | 11 (16) | 8 (37)
Decreased appetite (Metabolism and nutrition disorders) | 48 (68) | 35 (43)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (51) | 42 (81)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 26 (36)
Bone pain (Musculoskeletal and connective tissue disorders) | 16 (31) | 24 (34)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (28) | 25 (37)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 16 (22) | 15 (23)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 12 (15)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 9 (12) | 2 (4)
Spinal pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 9 (13)
Dizziness (Nervous system disorders) | 9 (11) | 9 (12)
Dysgeusia (Nervous system disorders) | 17 (26) | 13 (14)
Headache (Nervous system disorders) | 25 (35) | 30 (42)
Insomnia (Psychiatric disorders) | 15 (15) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (37) | 26 (40)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 17 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 14 (15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 16 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (10)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 (11) | 9 (31)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 14 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (18) | 14 (20)
Rash (Skin and subcutaneous tissue disorders) | 20 (29) | 30 (44)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (11) | 7 (14)
Hypertension (Vascular disorders) | 13 (22) | 7 (11)

LIMITATIONS AND CAVEATS:
Due to reassessment of the Primary Completion date (PCD) conditions, PCD was moved back to 22 January 2020. Interim survival data on patients transferring from this study to study 16996 (NCT02312960), as of analysis cutoff, was pooled with this study's data to increase the reliability of efficacy results. This pooling was specified in a supplemental SAP dated 24 Jun 2020. All other primary and secondary analysis details were specified in the main study SAP dated 14 Feb 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Where done for the purpose of filing a patent application, and where deemed necessary, the Sponsor/Bayer may request the PI of the Trial to postpone by 90 days the publication or presentation of a paper. The PI of the Trial may not publish the data yielded by its Site until all the results of the trial (in the case of a multi-center trial) have been published in their entirety or until at least 12 months have passed following completion, discontinuation or early termination of the Trial.

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT02258451/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT02258451/SAP_001.pdf